CLINICAL TRIAL: NCT04658498
Title: Improving Our Understanding of Respiratory Muscle Training to Facilitate Weaning From Mechanical Ventilation in the ICU
Acronym: TrainToWean
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Daniel Langer, PT, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S64871
Record Dates: First submitted 2020-11-18; First posted 2020-12-08 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Weaning Failure
Keywords: ICU acquired muscle weakness; IMT; Weaning outcomes; Maximal inspiratory pressure; Diaphragm EMG; Surface EMG; Diaphragm ultrasounds; Microbiopsies; Difficult to wean patients; Respiratory muscles

STUDY DESIGN:
Intervention Model Description: Double-blind, three arms parallel group randomized controlled trial with 1:1:1 allocation ratio
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (UC) (Experimental): Intermittent spontaneous breathing periods
  Interventions: Other: Procedure: Usual Care (UC)
- UC + High-intensity inspiratory muscle training (HI-IMT) (Experimental)
  Interventions: Other: Procedure: UC + HI-IMT
- UC + Low-intensity inspiratory muscle training (LI-IMT) (sham IMT) (Experimental)
  Interventions: Other: Procedure: UC + LI-IMT (sham IMT)

INTERVENTIONS:
Other: Procedure: Usual Care (UC) — Intermittent spontaneous breathing periods
  Arms: Usual Care (UC)
Other: Procedure: UC + HI-IMT — UC + Supervised daily sessions of training including 4 sets of 6-10 full vital capacity breaths against an external load using a tapered flow resistive device (POWERbreathe KH2, HaB International, UK). The maximum tolerable resistance allowing patients to inhale at least 70% of their inspiratory vital capacity will be chosen and progressively increased throughout the training period.
  Arms: UC + High-intensity inspiratory muscle training (HI-IMT)
Other: Procedure: UC + LI-IMT (sham IMT) — UC + superrvised daily sessions of training including 4 sets of 6-10 breaths at the lowest external imposable load with the tapered flow resistive device (POWERbreathe KH2, HaB International, UK) (i.e. 3 cmH2O).
  Arms: UC + Low-intensity inspiratory muscle training (LI-IMT) (sham IMT)

SUMMARY:
Mechanical ventilation is a life-saving treatment frequently applied in intensive care unit (ICU). Nonetheless, by putting at rest the respiratory muscles, it can lead to respiratory muscle weakness and atrophy, which are accompanied by prolonged duration of mechanical ventilation, difficult weaning and increased ICU mortality. Despite a strong theoretical rationale and some evidence supporting the use of inspiratory muscle training (IMT) to address respiratory muscle weakness and atrophy, the optimal approach to IMT remains largely uncertain. In fact, mechanistic studies evaluating physiological adaptations that occur in respiratory muscles of mechanically ventilated patients in response to different training regimens have not been conducted so far.

The aim of this study is to comprehensively investigate changes in respiratory muscle function in response to three different conditions that patients will be exposed to during their period of weaning from mechanical ventilation.

DETAILED DESCRIPTION:
A majority of mechanically ventilated patients develop respiratory muscle weakness during critical illness.

The potential value of implementing rehabilitative interventions for respiratory muscle conditioning are supported by observations showing that respiratory muscle weakness is associated with prolonged duration of mechanical ventilation, difficult weaning, and increased ICU mortality.

Despite a strong theoretical rationale and some evidence supporting its use, mechanistic studies evaluating physiological adaptations that occur in respiratory muscles of mechanically ventilated patients in response to different training regimens have not been performed so far. Consequently, the characterization of IMT modalities and of the optimal approach to IMT remain largely uncertain.

To date, the great part of the studies on the topic employed an external mechanical threshold device to perform trainings, in general adopting loads ranging between 10-50% of maximal inspiratory strength (i.e. maximal inspiratory pressure (PImax)). Intermittent spontaneous breathing periods (e.g. using partially assisted or spontaneous modes of ventilation) are also frequently applied as an activating stimulus to the respiratory muscles during periods of mechanical ventilation.

A tapered flow resistive load (TFRL) device (POWERbreathe KH2, HaB International, UK) has been already tested and implemented at University Hospital Leuven as a way of loading respiratory muscles in ICU patients. The TFRL approach represents a potential more optimal way of loading the respiratory muscles in patients on prolonged mechanical ventilation. Such a loading approach allows higher inspiratory tidal volumes to be reached and higher work and power generation during trainings, by adapting to changes in length-tension characteristics of the inspiratory muscles during inspiration.

With regards to training modalities, high-intensity IMT modalities by applying loads ranging between 30 and 50 %PImax, have not yet been proven to be associated with better improvements in respiratory muscle strength compared to low-intensity (sham) IMT modalities at loads not exceeding 10 %PImax.

On the other hand, no studies are available that assessed changes in respiratory muscle function beyond assessments of respiratory muscle strength in response to training.

Additionally, no training studies have tried to quantify the intrinsic loading of the patients (i.e. elastic and resistive resistances of the chest wall and the lungs) that muscles are exposed to in between periods of additional loading applied during IMT sessions.

The aim of this study is to comprehensively investigate changes in respiratory muscle function in response to three different conditions that difficult to wean patients will be exposed to during their weaning period. The complementary quantification of the entity of loading that respiratory muscles are bearing during assisted, spontaneous and resistive breathing would provide important novel insights on the optimization of IMT stimulus in different patients on prolonged mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Difficult and prolonged weaning patients
* Adequate oxygenation
* Febrile temperature < 38ºC
* Hemodynamic stability
* Stable blood pressure
* No or minimal vasopressors
* No myocardial ischemia
* Adequate hemoglobin and mentation
* Resolution of disease acute phase
* Able to follow simple verbal commands related to IMT
* Mechanically ventilated via a tracheostomy or endotracheal tube

Exclusion Criteria:

* Pre-existing neuromuscular disease
* Agitation
* Hemodynamically instable (arrhythmia, decompensated heart failure, coronary insufficiency)
* Hemoptysis
* Diaphoresis
* Spinal cord injury above T8
* Use of any type of home MV support prior to hospitalization
* Skeletal pathology that impairs chest wall movements
* Poor general prognosis or fatal outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (PImax) | Maximal duration of IMT treatment: 28 days
  Using a unidirectional valve which will be connected to the patient's tracheostomy tube or endotracheal tube for an uninterrupted period of 25 seconds.

SECONDARY OUTCOMES:
Diaphragm mobility, thickness and thickening fraction by ultrasounds | Maximal duration of IMT treatment: 28 days
  Assessment by diaphragm ultrasounds
Change in contractile material and structural alteration of sternocleidomastoid muscle | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies using Hematoxylin & Eosin (H&E) staining.
Change in fiber proportion of sternocleidomastoid muscle fibers | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies with immunostaining of the myosin heavy chain.
Change in size of sternocleidomastoid muscle fibers | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies with immunostaining of the myosin heavy chain.
Change in amount of satellite cells of sternocleidomastoid muscle | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies with Pax7 immunostaining
Change in amount of fibrotic tissue of sternocleidomastoid muscle | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies with Masson staining
Change of gene expression of atrophy/hypertrophy related pathways of sternocleidomastoid muscle | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies with RT2 profiler PCR array skeletal muscle, Qiagen
Change in cell proliferation of sternocleidomastoid muscle | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies cell proliferation assays
Change in cell differentiation of sternocleidomastoid muscle | Maximal duration of IMT treatment: 28 days
  By analyzing muscle microbiopsies cell differentiation assays
Change in Blood Flow Index (BFI) of extra-diaphragmatic respiratory muscles | Maximal duration of IMT treatment: 28 days
  Measured by near-infrared spectroscopy in combination with injections of the tracer indocyanine green dye (ICG), with optodes transcutaneously positioned on the scalene, sternocleidomastoid and upper rectus abdominis muscles.
Change in Tissue Oxygenation Index (TOI) of ex of extra-diaphragmatic respiratory muscles | Maximal duration of IMT treatment: 28 days
  Measured by near-infrared spectroscopy with optodes transcutaneously positioned on the scalene, sternocleidomastoid and upper rectus abdominis muscles
Change in signal amplitude of diaphragm electromyography | Maximal duration of IMT treatment: 28 days
  Diaphragm electromyography will be collected with an esophageal electrode catheter
Change in signal amplitude of electromyography of extra-diaphragmatic respiratory muscles | Maximal duration of IMT treatment: 28 days
  Electromyography of scalene, sternocleidomastoid, parasternal intercostal and rectus abdominis muscles will be collected through surface electromyography electrodes
Esophageal and gastric pressure | Maximal duration of IMT treatment: 28 days
  Using a multifunction nasogastric catheter

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dres M, Goligher EC, Heunks LMA, Brochard LJ. Critical illness-associated diaphragm weakness. Intensive Care Med. 2017 Oct;43(10):1441-1452. doi: 10.1007/s00134-017-4928-4. Epub 2017 Sep 15. PMID 28917004
- [Background] Vorona S, Sabatini U, Al-Maqbali S, Bertoni M, Dres M, Bissett B, Van Haren F, Martin AD, Urrea C, Brace D, Parotto M, Herridge MS, Adhikari NKJ, Fan E, Melo LT, Reid WD, Brochard LJ, Ferguson ND, Goligher EC. Inspiratory Muscle Rehabilitation in Critically Ill Adults. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2018 Jun;15(6):735-744. doi: 10.1513/AnnalsATS.201712-961OC. PMID 29584447
- [Background] Supinski GS, Callahan LA. Diaphragm weakness in mechanically ventilated critically ill patients. Crit Care. 2013 Jun 20;17(3):R120. doi: 10.1186/cc12792. PMID 23786764
- [Background] Dres M, Goligher EC, Dube BP, Morawiec E, Dangers L, Reuter D, Mayaux J, Similowski T, Demoule A. Diaphragm function and weaning from mechanical ventilation: an ultrasound and phrenic nerve stimulation clinical study. Ann Intensive Care. 2018 Apr 23;8(1):53. doi: 10.1186/s13613-018-0401-y. PMID 29687276
- [Background] Elkins M, Dentice R. Inspiratory muscle training facilitates weaning from mechanical ventilation among patients in the intensive care unit: a systematic review. J Physiother. 2015 Jul;61(3):125-34. doi: 10.1016/j.jphys.2015.05.016. Epub 2015 Jun 16. PMID 26092389
- [Background] Langer D, Charususin N, Jacome C, Hoffman M, McConnell A, Decramer M, Gosselink R. Efficacy of a Novel Method for Inspiratory Muscle Training in People With Chronic Obstructive Pulmonary Disease. Phys Ther. 2015 Sep;95(9):1264-73. doi: 10.2522/ptj.20140245. Epub 2015 Apr 9. PMID 25858974
- [Background] Hoffman M, Van Hollebeke M, Clerckx B, Muller J, Louvaris Z, Gosselink R, Hermans G, Langer D. Can inspiratory muscle training improve weaning outcomes in difficult to wean patients? A protocol for a randomised controlled trial (IMweanT study). BMJ Open. 2018 Jun 30;8(6):e021091. doi: 10.1136/bmjopen-2017-021091. PMID 29961023
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Derived] Poddighe D, Van Hollebeke M, Clerckx B, Janssens L, Molenberghs G, Van Dyck L, Muller J, Gunst J, Meersseman P, Peetermans M, Hermans G, Gosselink R, Langer D. Inspiratory effort and respiratory muscle activation during different breathing conditions in patients with weaning difficulties: An exploratory study. Aust Crit Care. 2025 May;38(3):101152. doi: 10.1016/j.aucc.2024.101152. Epub 2025 Jan 21. PMID 39842329